CLINICAL TRIAL: NCT06184386
Title: Efficiency of Parental Feeding Support to Strengthen NIDCAP and Favor Eating Development in Preterm Newborns as Compared With a Retrospective Orofacial Stimulation Standardized and Routine Clinical Practice
Brief Title: Oral Feeding Delay Prevention in Preterm Newborns
Acronym: PARENTALIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 20-161
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Preventive Care
Keywords: preterm newborns; individualized developmental care; parental suppport for nursing; orofacial stimulations; oral feeding

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective NIDCAPARENTALIM: A group of prospectively assigned preterm newborns that will be included in NIDCAP strengthened with a practice focalized on feeding, named PARENTALIM.
  Interventions: Other: NIDCAPARENTALIM
- Retrospective SOFS: A group of retrospectively assigned preterm newborns that had standardized orofacial stimulations named SOFS.
  Interventions: Behavioral: SOFS

INTERVENTIONS:
Other: NIDCAPARENTALIM — PARENTALIM practice that strengthens the NIDCAP. It is proposed in a routine way in the NICU since 2019. PARENTALIM supports and monitors parental implication in nursing care. It is led by a speach language therapist specialized in early feeding development who proposes 5 individualized interviews and uses an educational booklet on eating development care with a lot of illustrations and few words.
  Groups: Prospective NIDCAPARENTALIM
Behavioral: SOFS — SOFS is a behavioral practice of orofacial stimulations. Il has been mainly carried out by nurses or a speach language therapist specialized in early feeding development. SOFS has been applied through routine protocol in the NICU until 2018.
  Groups: Retrospective SOFS

SUMMARY:
Preventing oral feeding delays in preterm newborns remains a stake for NICU nowadays. Indeed, it lengthens hospitalization duration, distorts parent-newborns relationships, and increases the risks of adverse nursing outcomes. Does a routine individualized developmental preventive feeding care implying parents favors earlier autonomous oral feeding achievement in preterm newborns as compared with a standardized routine program of orofacial stimulations, despite neonatal risks that every preterm newborn cumulates during hospitalization stay ?

DETAILED DESCRIPTION:
The goal of this observational study is to compare the efficiency of two routine preventive feeding care in preterm newborns, taking into account neonatal cumulated risks for each preterm newborn participant. The main question it aims to answer is: Does a prospective individualized routine developmental preventive feeding care leads to earlier oral feeding achievement in preterm newborns despite individual risks, as compared with a retrospective standardized routine program. The group of preterm newborns prospectively assigned in the study will be included in NIDCAP strengthen with a parental support on nursing care named PARENTALIM. The group of preterm newborns retrospectively assigned in the study received orofacial stimulations in a standardized protocol way (SOFS) Researchers will compare prospective and retrospective groups to see if the prospective group achieve autonomous oral feeding, despite individual neonatal cumulated risks, significantly earlier than retrospective group.

ELIGIBILITY:
Inclusion Criteria:

* Parents of preterm newborns born before 34 weeks of amenorrhea
* Parents who agree participating in the study after signing an informed consent.
* Minimal delay of 72 hours and maximal delay of 15 days after birth to inform parents and wait their consent.

Exclusion Criteria:

* Parents of preterm newborns born after 35 weeks of amenorrhea
* Parents who disagree participating in the study, even after signing the informed consent.
* Parents of preterm newborns born with cerebral, maxillo-facial, digestive, cardiac, genetic or syndromic abnormalities.

Ages: 3 Days to 10 Weeks | Sex: All
Age Groups: Child
Study Population: Preterm newborns born before 34 weeks of amenorrhea with variable but moderated neonatal risks and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
The precocity of autonomous oral feeding achievement taking into account the index of cumulated neonatal risks | 5 years
  The corrected age in ammenorhea weeks at which preterm newborn achieve autonomous oral feeding will be divided by the index of cumulated neonatal risks scored from the updated risk inventory initially proposed by Sheiner and Sexton in 1991

SECONDARY OUTCOMES:
The duration of oral feeding transition | 5 years
  The duration from the moment when preterm newborn takes 5 ml per kg per day and until the moment when autonomous oral feeding is achieved.

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTEL BLAISON, Principal Investigator — Speach language Therapist at University Hospital
Locations (1):
- Maryse Delaunay, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided